CLINICAL TRIAL: NCT05801913
Title: A Pilot / Feasibility Study of Autologous CMV-Specific CD19-CAR T Cells Plus CMV-MVA Triplex Vaccine in Patients With Intermediate or High Grade B-Lineage Non-Hodgkin Lymphoma
Brief Title: Genetically Modified T-cells (CMV-Specific CD19-CAR T-cells) Plus a Vaccine (CMV-MVA Triplex) for the Treatment of Intermediate or High Grade B-Cell Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22459; NCI-2023-02195 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22459 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: High Grade B-Cell Non-Hodgkin's Lymphoma; Intermediate Grade B-Cell Non-Hodgkin's Lymphoma; Recurrent B-Cell Non-Hodgkin Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Specimen Handling; Biopsy; Leukapheresis; Magnetic Resonance Spectroscopy; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CMV-specific CD19-CAR T cells, triplex vaccine) (Experimental): Patients undergo leukapheresis on day -30 and receive lymphodepleting chemotherapy on days -10 to -3 per SOC on study. Patients then receive CMV-specific CD19-CAR T cells IV on day 0 and CMV-MVA triplex vaccine IM on days 28 and 56 in the absence of unacceptable toxicity on study. Patients also undergo x-ray during screening and on study, as well as PET, CT, MRI, blood sample collection, and bone marrow biopsy on study and during follow-up.
  Interventions: Biological: Anti-CD19-CAR CMV-specific T-lymphocytes; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Leukapheresis; Procedure: Lymphodepletion Therapy; Procedure: Magnetic Resonance Imaging; Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine; Procedure: Positron Emission Tomography; Procedure: X-Ray Imaging

INTERVENTIONS:
Biological: Anti-CD19-CAR CMV-specific T-lymphocytes — Given IV
  Other Names: Anti-CD19-CAR CMV-specific T-cells; CMV-specific CD19 CAR-T Cells; CMV-specific CD19-CAR T Cells
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Leukapheresis — Undergo leukapheresis per SOC
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Procedure: Lymphodepletion Therapy — Undergo lymphodepletion chemotherapy per SOC
  Other Names: Lymphodepleting Therapy; Lymphodepletion
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine — Given IM
  Other Names: CMV-MVA Triplex Vaccine; Multi-antigen CMV-Modified Vaccinia Ankara Vaccine
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Procedure: X-Ray Imaging — Undergo x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase I trial studies the safety and feasibility of cytomegalovirus (CMV) specific CD19-chimeric antigen receptor (CAR) T cells in combination with the CMV-modified vaccinia Ankara (MVA) triplex vaccine following lymphodepletion in treating patients with intermediate or high grade B-cell non-Hodgkin lymphoma (NHL) that has come back after a period of improvement (relapsed) or that does not respond to treatment (refectory). CAR T cells are a type of treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein on the patient's cancer cells is added in the laboratory. The special receptor is called CAR. Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion. Vaccines such as CMV-MVA triplex are made from gene-modified viruses and may help the body build an effective immune response to kill cancer cells. Giving CMV-specific CD19-CAR T-cells plus the CMV-MVA triplex vaccine may help prevent the cancer from coming back.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the safety and describe the toxicity profile of anti-CD19-CAR CMV-specific T-lymphocytes (CMV-specific CD19-CAR T cells) as monotherapy and when given in combination with a multi-peptide CMV-modified vaccinia Ankara vaccine (CMV-MVA Triplex) following standard of care lymphodepletion.

SECONDARY OBJECTIVES:

I. Determine the feasibility of autologous CMV-specific CD19-CAR T cell manufacturing, as assessed by the ability to meet the required cell dose and product release requirements.

II. Estimate the overall and complete disease response rate at days 28 and 84 after CAR T cell infusion.

III. Determine short- and longer-term CMV-specific CD19-CAR T cell in vivo expansion and persistence.

IV. Assess whether the CMV-specific CD19-CAR T cells respond to CMV-MVA Triplex vaccine.

V. Estimate the rate of CMV reactivation after CAR T cell. VI. Estimate the one-year progression-free survival (PFS) rate and median overall survival (OS) post-CAR T cell infusion.

EXPLORATORY OBJECTIVE:

I. Assess whether the CMV-specific CD19-CAR T cells respond to CMV-MVA Triplex vaccine when administered to participants that received CAR T cells only in the safety lead-in portion in the expansion phased of the study (i.e., once safety of the CMV-MVA Triplex vaccine is established in the feasibility portion of the study).

OUTLINE: This is a dose-escalation study of CMV-specific CD19-CAR T cells followed by a dose-expansion study.

Patients undergo leukapheresis on day -30 and receive lymphodepleting chemotherapy on days -10 to -3 per standard of care (SOC) on study. Patients then receive CMV-specific CD19-CAR T cells intravenously (IV) on day 0 and CMV-MVA triplex vaccine intramuscularly (IM) on days 28 and 56 in the absence of unacceptable toxicity on study. Patients also undergo x-ray during screening and on study, as well as positron emission tomography (PET), computed tomography (CT), magnetic resonance imaging (MRI), blood sample collection, and bone marrow biopsy on study and during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Note: For research participants who do not speak English, a short form consent may be used with a City of Hope (COH) certified interpreter/translator to proceed with screening and leukapheresis, while the request for a translated full consent is processed
* Age: >= 18 years
* Karnofsky Performance Status (KPS) >= 70
* Life expectancy >= 16 weeks at the time of enrollment
* Patients requiring treatment for relapsed or refractory intermediate or high-grade B cell NHL (e.g., diffuse large B-cell lymphoma [DLBCL], mantle cell lymphoma [MCL], or transformed NHL) who are not eligible for, or who refuse, or have previously received autologous hematopoietic cell transplantation (autoHCT)

  * Note: COH pathology review should confirm that research participant's diagnostic material is consistent with history of intermediate or high-grade CD19+ malignancy
* No known contraindications to leukapheresis, lymphodepleting chemotherapy, steroids or tocilizumab, smallpox vaccine and any other MVA-based vaccines
* Patient must be CMV seropositive
* Total serum bilirubin =< 2.0 mg/dL
* Participants with Gilbert syndrome may be included if their total bilirubin is =< 3.0
* Aspartate aminotransferase (AST) < 2.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) < 2.5 x ULN
* Serum creatinine =< 2.5 x ULN or estimated creatinine clearance of >= 40 mL/min per the Cockcroft-Gault formula, and the participant is not on hemodialysis
* Absolute neutrophil count >= 1000/uL (Transfusions and growth factors must not be used to meet these requirements at initial screening)
* Hemoglobin (Hb) >= 8 g/dl (Transfusions and growth factors must not be used to meet these requirements at initial screening)
* Platelet count >= 50,000/uL (>= 30,000/uL if bone marrow plasma cells are >= 50% of cellularity) (Transfusions and growth factors must not be used to meet these requirements at initial screening)
* Left ventricular ejection fraction >= 45% within 8 weeks before enrollment
* Oxygen (O2) saturation > 92% without requiring supplemental oxygen
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Prior allogeneic stem cell transplant unless the participant has recovered from transplantation and does not have active graft versus host disease (GVHD)
* Growth factors within 14 days of enrollment
* Platelet transfusions within 7 days of enrollment
* Concurrent use of systemic steroids or chronic use of immunosuppressant medications. Recent or current use of inhaled or topical steroids in standard doses is not exclusionary. Physiologic replacement of steroids (prednisone =< 5 mg/day, or equivalent doses of other corticosteroids) is allowed
* Patients with active autoimmune disease requiring systemic immune suppressive therapy are not allowed
* Participants may not be receiving any other investigational agents or concurrent biological therapy, chemotherapy, or radiation therapy
* Any standard contraindications to lymphodepleting chemotherapy and/or CAR T-cell therapy per standard of care practices at COH
* Subjects with clinically significant arrhythmia or arrhythmias not stable on medical management within two weeks of screening
* Subjects with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system (CNS), including seizure disorder, any measurable masses of CNS, or any other active CNS disease

  * Note: Research participants with a history of CNS disease that has been effectively treated to complete remission (< 5 white blood cell [WBC]/mm^3 and no blasts in cerebral spinal fluid [CSF]) will be eligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents or cetuximab
* Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia
* History of stroke or intracranial hemorrhage within 6 months prior to screening
* History of other malignancies, except for malignancy surgically resected (or treated with other modalities) with curative intent, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; non-muscle invasive bladder cancer; malignancy treated with curative intent with no known active disease present for >= 3 years
* Clinically significant uncontrolled illness
* Active infection requiring antibiotics
* Immunodeficiency virus (human immunodeficiency virus [HIV]) positive
* Active viral hepatitis
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity | Up to 28 days
  Toxicities will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0, and the revised American Society for Transplantation and Cellular Therapy (ASTCT) cytokine release syndrome (CRS) grading systems. Will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome.
Incidence of adverse events | Up to 15 years
  Will be assessed and graded according to the NCI CTCAE v5.0, and the ASTCT consensus grading for CRS and neurotoxicity associated with immune effector cells.

SECONDARY OUTCOMES:
Feasibility as assessed by the ability to meet the required cell dose and product release requirement | Up to 56 days
  Feasibility will be assessed by achieving the proposed dose of CMV-specific CD19-CAR T cells per product and meeting product release requirements for enrolled participants. The goal is to manufacture 10 x 10^6 cells (this is a flat dose).
Short- and long-term cytomegalovirus (CMV)-specific CD19-chimeric antigen receptor (CAR) T cell expansion and persistence | Up to 15 years
  Will be assessed longitudinally. Persistence is defined as detection of >= 0.1% of CMV-specific CD19-CAR T cells in CD3+ cells in peripheral blood, 28 days after vaccine administration, by flow cytometry and Woodchuck Hepatitis Virus Posttranscriptional Regulatory Element quantitative polymerase chain reaction (Q-PCR). Expansion is defined as an increase of 2-fold in CMV-specific CD19-CAR T cells after Triplex administration compared with pre-vaccination cell number. Response to Triplex will be assessed based on numbers of EGFR+, pp65-specific interferon gamma (IFNy)+ and CD137+T cells.
Clinically significant CMV reactivation | Up to 15 years
  Clinically significant defined as > 1250 IU/ml or 500 GC/mL) CMV reactivation requiring management treatment after CAR T cell infusion as assessed by PCR.
Disease response (complete response/minor response/partial response/disease progression/stable disease) | 28 and 84 days after CAR T cell infusion
  Will be assessed according to International Working Group consensus response evaluation criteria in lymphoma 2017. The specific time trend for CMV-specific CD19-CAR T cells will be assessed using linear mixed effects modeling. The overall fit of the model will be evaluated graphically by taking a scatter plot of data for the CAR T cells and applying an overlay of the line generated by the model. To assess changes over time, functional regression modeling will be used.
Progression-free survival | Time from the start of lymphodepletion to the time of disease relapse, progression or death, whichever occurs first, assessed at 1 year and up to 15 years
  Will be estimated using the product-limit method of Kaplan and Meier.
Overall survival | Time from the start of lymphodepletion to death, assessed up to 15 years
  Will be estimated using the product-limit method of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie L Popplewell, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States